CLINICAL TRIAL: NCT06586073
Title: Evaluation of the Efficacy of Topical Cosmetic Products in Patients with Hand and Foot Syndrome (HFS) Undergoing Oncological Treatments
Brief Title: Topical Cosmetic Products for Hand and Foot Syndrome
Status: Completed | Type: Observational
Sponsor: Dermophisiologique s.r.l (Industry)
Collaborators: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: R1633/22-IEO 1748
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Hand Foot Skin Syndrome
Keywords: Hand-foot syndrome; skin toxicity; cancer treatments; quality of life; cosmetic products
MeSH Terms: conditions — Hand-Foot Syndrome | interventions — Cosmetics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 45 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Diagnosed cancer patients receiving different therapies with hand-foot syndrome skin side effects: Participants were diagnosed cancer patients receiving chemotherapy and targeted or hormonal treatments. Recruitment was performed by the medical oncologists based on the presence of Hand-foot syndrome (HFS) grade 1 symptoms. The severity of HFS was graded according to the The National Cancer Institute-Common Terminology Criteria for Adverse Events Criteria (NCI-CTCAE) version 5.0. All patients enrolled were provided with a kit of four cosmetic products formulated explicitly for cancer skincare
  Interventions: Other: cosmetic products

INTERVENTIONS:
Other: cosmetic products — All patients enrolled were prescribed four cosmetic products (Ontherapy® by Dermophisiologique) for skin treatment: a cleansing cream, a soothing and nourishing cream, an anti-desquamation cream with urea 5%, and an emollient mixture. Patients were instructed to use each product at home for 45 days, following a specific protocol: in the morning, apply the affinity cleansing cream during skin cleansing, followed by the anti-desquamation cream, while in the evening, apply affinity cleansing cream followed by the application of the emollient mixture and then the soothing and nourishing cream.

SUMMARY:
The aim of the study is to evaluate the efficacy of a dermocosmetic protocol in reducing the main cutaneous side effects that occur in palmar-plantar erythrodysesthesia syndrome in subjects with a tumor diagnosis, undergoing chemotherapy and targeted treatments such as target therapy and radiotherapy.

DETAILED DESCRIPTION:
Cancer patients undergoing active oncological treatment (chemotherapy, biological therapies, radiotherapy) experience multiple side effects, including skin toxicity, which negatively affects their quality of life, increasing the risk of interrupting cancer therapy. Symptomatic therapy is often neglected and prescribed late in the course of the disease. Many patients undergoing anti-cancer therapies experience adverse skin reactions such as dry skin, rashes, redness, and itching. Dry skin, erythema, and nail lesions are particularly common for those undergoing chemotherapy and targeted treatments such as target therapy and radiotherapy.

Cleansing must be done by affinity, that is, with an emulsification mechanism and not solubilization, through the use of "sebum-like" fatty substances to remove only the excess lipids on the skin surface and the dirt attached to them. This eudermic cleansing without the use of surfactants does not solubilize the epidermal lipids that are fundamental in the structure of the hydrolipidic film, maintaining the right protection and hydration of the skin.

Therefore, the main objective of the following study is to evaluate the efficacy of 4 topical cosmetic products specifically formulated for patients undergoing oncological therapy in the management of palmar-plantar erythrodysesthesia syndrome, a skin toxicity typical of oncological treatments, which causes skin alterations such as erythema and/or xerosis and/or mild to moderate nail damage, to ensure an improvement of the skin condition during therapy.

ELIGIBILITY:
Inclusion Criteria:

* Cancer diagnosis undergoing oncological therapy with chemotherapeutic agents, targeted therapy, immunotherapy hormonal treatments
* Patients with grade 1 of Hand-foot syndrome (HFS) Male and female patients 18 age or more
* Conditions favoring the correct execution of the proposed program
* Signature of informed consent, privacy and the form for the use of the data

Exclusion Criteria:

* Pregnancy or breastfeeding in progress
* Other skin toxixities different from HFS
* Patients with HFS adverse skin symptoms higher than grade 1
* Psychic or other disorderes
* Patients with preexisting skin disorders thet could interfere with thw study results (like dermatitis, prosriais)
* Known hypersensitivity or allergy to one of the components of the products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants were diagnosed cancer patients recruited from the oncology departments at the European Institute of Oncology, Milan, Italy.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the mean skin hydration index at 45 days | Baseline and 45 days
  Changes from the baseline of skin hydration were assessed using a Corneometer® CM 825 probe that analyze water related changes in the skin's electrical capacitance. All measurements reported are the average of three assessments obtained on two skin areas: the right hand 's dorsum and the right foot's dorsum

SECONDARY OUTCOMES:
Change from Baseline in the mean skin redness index at 45 days | Baseline and 45 days
  Changes from the baseline of skin redness (erythema) were measured photometrically by a Mexameter ® MX 18 30 32 All measurements reported are the average of three assessments obtained on four skin areas: the palm of the right hand, fingertip of the right hand, sole of the right foot and fingertip of the right foot.
Change from Baseline in the mean overall Skindex-16 score at 45 days | Baseline and 45 days
  The impact of skin manifestations on patient Quality of life (QoL) was evaluated using the Skindex 16, a 16 item self report questionnaire. It is composed of three subscales: perceived symptoms (items 1-5), emotions (items 6-11), and daily functions (items 12-16).Responses to each item were transformed into a linear scale of 100, varying from 0 (never bothered) to 100 (corresponding to 6, always bothered). Each raw score was then normalized for the statistical to 100 (corresponding to 6, always bothered). Each raw score was then normalized for the statistical analysis. The final score is the average of the patient's responses in each domain.
Assessment from baseline of compliance with the study protocol at 45 days | Baseline and 45 days
  The compliance of patients with the product use protocol was assessed through a specific diary within 45 days, divided into morning and evening, containing two boxes to tick (YES for products applied or NO for products not applied). Additionally, there is a NOTES section where the patient can input the reason for not applying the product
Change in the degree of toxicity of hand-foot syndrome using the v5.0 scale of the National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE). | Baseline and 45 days
  The oncologist and dermatologist clinically evaluated HFS severity by comparing patient pictures taken standardized at baseline and at the end of the study (45 days) on four body areas: the back of the hand, the back of the foot, the palm, and the sole. The oncologist assessed the change in the degree of hand-foot syndrome toxicity using the National Cancer Institute -Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0 scale. The dermatologist used a three-point evaluation (improvement, stability, worsening) to assess the change in HFS-related skin symptoms (erythema, xerosis, and desquamation). Treatment benefit was evaluated according to the reduction of the NCI CTCAE grade and the improvement of skin symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Ida Minchella, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology (IEO), Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Biswal SG, Mehta RD. Cutaneous Adverse Reactions of Chemotherapy in Cancer Patients: A Clinicoepidemiological Study. Indian J Dermatol. 2018 Jan-Feb;63(1):41-46. doi: 10.4103/ijd.IJD_65_17. PMID 29527024
- [Background] Saadet ED, Tek I. Evaluation of chemotherapy-induced cutaneous side effects in cancer patients. Int J Dermatol. 2022 Dec;61(12):1519-1526. doi: 10.1111/ijd.16361. Epub 2022 Jul 22. PMID 35867950